CLINICAL TRIAL: NCT03105869
Title: Repeatability of Positron Emission Tomography (TEP) With fluorométhyl-(18F)-diméthyl-2-hydroxyéthyl-ammonium
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RECHOL
Record Dates: First submitted 2017-04-04; First posted 2017-04-10 (Actual); Last update posted 2017-06-26 (Actual); Status verified 2017-06

CONDITIONS: Prostate Cancer
Keywords: repeatability; positron emission tomography (PET); fluorocholine
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: test and retest in a single group of patient
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- fluorocholine PET/CT (Experimental): all patients will undergo a second PET/CT with fluorocholine
  Interventions: Diagnostic Test: fluorocholine PET/CT

INTERVENTIONS:
Diagnostic Test: fluorocholine PET/CT — standard diagnostic PET/CT procedure

SUMMARY:
Monocentric study. Objective : Determination of the repeatability of fluorocholine PET/CT in prostate cancer

DETAILED DESCRIPTION:
A second PET/CT with fluorocholine is performed within 2 weeks after a first examination performed in patient referred for an initial prostate cancer or a biological suspicion of relapse.

ELIGIBILITY:
Inclusion criteria :

* biological suspicion of relapse of prostate cancer or initial staging of prostate cancer
* positive PET/CT with fluororocholine

Exclusion criteria :

-none

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — male
Enrollment: 20 (Actual)
Dates: Start 2014-12-16 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
reproducibility of the results | 2 weeks
  Comparison of the number and location of identified lesions and comparison of lesion uptake

CONTACTS AND LOCATIONS:
Overall Officials: Catherine CHEZE LE REST, Principal Investigator — CHU Poitiers

IPD SHARING:
Plan to Share IPD: No